CLINICAL TRIAL: NCT06021860
Title: A Phase IV, Two-part, Open-label Study Assessing the Pharmacokinetics, Safety and Pharmacodynamics of Single and Multiple Doses of Spironolactone Oral Suspension in Pediatric Patients With Edema Due to Heart Failure or Cirrhosis
Brief Title: A Phase IV, Two-part, Open-label Study Assessing the Pharmacokinetics, Safety and Pharmacodynamics of Spironolactone Oral Suspension in Pediatric Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CMP Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREA 3256-4
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Edema Due to Heart Failure or Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Canrenoic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1: multiple doses spironolactone oral suspension (Group 1) (Experimental): Patients aged ≥12 to ≤17 years of age in Part 1 of the study, administered spironolactone oral suspension QD for 10 days
  Interventions: Drug: Spironolactone Oral Suspension
- Part 1: multiple doses spironolactone oral suspension (Group 2) (Experimental): Patients aged ≥6 to <12 years of age in Part 1 of the study, administered spironolactone oral suspension QD for 10 days
  Interventions: Drug: Spironolactone Oral Suspension
- Part 1: multiple doses spironolactone oral suspension (Group 3) (Experimental): Patients aged ≥2 to <6 years of age in Part 1 of the study, administered spironolactone oral suspension QD for 10 days
  Interventions: Drug: Spironolactone Oral Suspension
- Part 1: single and multiple doses spironolactone oral suspension (Group 4) (Experimental): Patients aged from birth to <2 years of age in Part 1 of the study, administered spironolactone oral suspension as a single dose, and then QD for 10 days
  Interventions: Drug: Spironolactone Oral Suspension
- Part 2: multiple doses spironolactone oral suspension (Group 1) (Experimental): Patients aged ≥12 to ≤17 years of age in Part 2 of the study, administered low or high dose spironolactone oral suspension QD for 10 days
  Interventions: Drug: Spironolactone Oral Suspension
- Part 2: multiple doses spironolactone oral suspension (Group 2) (Experimental): Patients aged ≥6 to ≤12 years of age in Part 2 of the study, administered low of high dose spironolactone oral suspension QD for 10 days
  Interventions: Drug: Spironolactone Oral Suspension
- Part 2: multiple doses spironolactone oral suspension (Group 3) (Experimental): Patients aged ≥2 to ≤6 years of age in Part 2 of the study, administered low or high dose spironolactone oral suspension QD for 10 days
  Interventions: Drug: Spironolactone Oral Suspension
- Part 2: single and multiple doses spironolactone oral suspension (Group 4) (Experimental): Patients aged from birth to <2 years of age in Part 2 of the study, administered low or high dose spironolactone oral suspension as a single dose, and then QD for 10 days
  Interventions: Drug: Spironolactone Oral Suspension

INTERVENTIONS:
Drug: Spironolactone Oral Suspension — Spironolactone will be dosed on a mg/kg basis, with actual weight on Day 1 (pre-dose) determining the spironolactone suspension volume administered. Therefore, for a given patient, the dose administered on Day 1, based on the weight measured on Day 1, will be administered throughout their participation in the study.
  Spironolactone will be administered as a single dose in the single-dose periods (Group 4, Parts 1 and 2), and as QD dosing in the multiple-dose periods (Groups 1 to 4, Parts 1 and 2).
  The low and high doses to be administered during Part 2 of the study will be determined by the Safety Review Committee following their review of Part 1 data.
  Other Names: Carospir®

SUMMARY:
This is a 2-part, 2 periods per part, open-label study with spironolactone oral suspension in pediatric patients with edema due to HF or hepatic cirrhosis. Both study parts will evaluate the safety, PK and PD of multiple doses of spironolactone in patients aged from birth to ≤17 years of age.

DETAILED DESCRIPTION:
This is a 2-part, 2 periods per part, open-label study with spironolactone oral suspension in pediatric patients with edema due to heart failure or hepatic cirrhosis. Both study parts will evaluate the safety, PK and PD of multiple doses of spironolactone. In Part 1 of the study, a single dose of spironolactone oral suspension will be administered. In Part 2 of the study, a low and a high dose of spironolactone oral suspension will be selected based on the results of Part 1, and will be administered to patients.

Part 1 During a 14-day screening period, 18 patients will be enrolled in parallel to 1 of 3 groups, with 6 patients in each group (Group 1: adolescents: ≥12 to ≤17 years of age; Group 2: children: ≥6 to <12 years of age; and Group 3: children: ≥2 to <6 years of age). For these patients the study will begin with a multiple-dose period, where patients will be administered a once-daily (QD) 1.5 mg/kg dose of spironolactone oral suspension for a total of 10 days. There will then be a 30-day follow-up period. Following the conclusion of Groups 1 though 3 in the multiple-dose period of Part 1 of the study, a Safety Review Committee will review all data from Groups 1 though 3 and determine whether and how the study should proceed. If the study proceeds as planned, 6 patients aged from birth to <2 years of age will be enrolled into Group 4 during a 14-day screening period. These patients will begin the study with a single-dose period, during which they will be administered a single dose of spironolactone oral suspension at a dose determined by the Safety Review Committee. They will be followed for 7 days. They will proceed into the multiple-dose period, and will be administered a QD dose (at the same level received in the single-dose period), for a total of 10 days. There will then be a 30-day follow-up period.

Part 2 After reviewing data from Part 1 of the study, the Safety Review Committee will make the decision whether to open enrollment in Part 2 of the study, whether to open enrollment to all age groups, and the low and high doses of spironolactone oral suspension to be used. If the study proceeds as planned, 54 patients will be enrolled in parallel to either Group 1, 2, or 3, with 18 patients in each. Nine patients in each group will be assigned a low dose of spironolactone oral suspension, and 9 patients will be assigned to a high dose. These patients will proceed as described in Part 1, with a multiple-dose period where spironolactone oral suspension is administered QD at either a low or high dose for a total of 10 days, followed by a 30-day follow-up period. Following the conclusion of Groups 1 through 3 in the multiple-dose period of Part 2, eighteen patients aged from birth to <2 years of age will be enrolled into Group 4. Nine patients will be assigned to a low dose of spironolactone oral suspension, and 9 patients will be assigned to a high dose. As described for Part 1, these patients will begin the study with a single-dose period during which they will be administered a single dose (low or high) of spironolactone oral suspension and then followed for 7 days before being administered a QD dose (at the same level received in the single-dose period), for a total of 10 days. There will then be a 30-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patient or patient's parent or legal guardian (if applicable) provides written consent to participate in the study and provides written informed consent prior to any study procedures being performed.
* Female patients of childbearing potential may be enrolled if they are practicing abstinence and have a negative urine pregnancy test at Screening and/or Day 1, or using 2 forms of highly effective contraception.
* Male patients with female partners of childbearing potential may be enrolled if they are practicing abstinence or using 2 forms of highly effective contraception.
* Patients must agree to stay in clinic or the supervised care unit on specified days.
* Patients must have past diagnosis of edema (includes peripheral and/or pulmonary edema) due to heart failure or hepatic cirrhosis requiring, or expected to require, treatment with spironolactone in the investigator's judgment.
* Stable therapy for chronic comorbidities (unrelated to HF or cirrhosis, and as approved by the Investigator and Medical Monitor) is allowed, with no changes to these medications in the 72 hours prior to administration of study drug on Day 1 and for the duration of the study.
* Loop diuretics (such as furosemide), if taken, must be stable for 72 hours prior to dosing of spironolactone on Day 1 and to the extent possible for the remainder of the study.

Exclusion Criteria:

* Prematurity, defined as babies not born out of full-term pregnancy (Group 4 only) (˂38 weeks of gestation).
* Have received spironolactone or eplerenone in the past 14 days before Screening.
* Current acute renal injury (as determined by the Investigator).
* Chronic renal insufficiency: estimated glomerular filtration rate calculated using the modified Schwartz formula <30% of expected for age and size.
* Electrocardiogram corrected QT interval of >460 msec.
* Patients who have received blood transfusions within 2 weeks prior to Screening, and for the duration of treatment.
* Electrolyte disturbances (at Screening):
* Has poorly controlled diabetes (HbA1c >8.5%).
* Requires circulatory assistance device.
* Any prior solid organ transplant.
* Major surgery (as determined in the Investigator's judgement) within 1 month of dosing unless approved by the investigator and medical monitor.
* Has known history of hypersensitivity or intolerance to spironolactone or other ingredients in the study drug formulation.
* Has known contraindication to treatment with spironolactone.
* Requires treatment with a medication known to affect spironolactone exposure as indicated in the contraindications and drug interaction recommendations listed in the label.
* Is pregnant or lactating.
* Participation in a drug study or exposure to any other investigational drug or placebo within 2 months of study drug administration in the current study.
* Use of thiazide diuretics, K-sparing diuretics, any hormonal contraceptive agent, or consumption of any nutrients known to modulate the activity of CYP450 enzymes outside of the permitted use.
* Concomitant prescription medications outside the stable standard of care regimen for edematous conditions and other chronic comorbidities administered within 2 weeks prior to study drug administration.
* Patients who have smoked or used smoking-cessation or nicotine-containing products within 3 months of the first dose of the study drug until last/End of Study Visit.
* Consumption of caffeine, energy drinks, alcohol, or recreational drugs (including marijuana) within 72 hours prior to administration of study drug on Day 1 and for the duration of the study.
* Uncontrolled (with treatment), active bacterial, fungal, or viral infections within 72 hours prior to Screening.
* Screening laboratory tests positive for HIV, hepatitis B, and hepatitis C.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Part 1: Absorption rate constant (Ka) of spironolactone (time^-1) in the multiple-dose period | Pre-dose (Day 1) to 22-26 hours post-dose (Day 11)
  Patients will be assigned to a pharmacokinetic sampling schedule as follows:
  Group 1, Subgroup 1 - Day 1: pre-dose; Day 10; 0.08-0.5 hours, 1-1.5 hours, 2-3 hours, 4-6 hours, 10-13 hours post-dose; Day 11: 22-26 hours post-dose
  Group 1, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.5-1 hour, 1.5-2 hours, 3-4 hours, 6-8 hours post-dose; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 1 - Day 1: pre-dose; Day 10: 0.08-0.75 hours, 1.5-2.5 hours, 3.5-6 hours, 10-13 hours; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.75-1.5 hours, 2.5-3.5 hours, 6-8 hours, 10-13 hours post-dose
  Group 4: the pharmacokinetic sampling schedule during the multiple-dose period for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3.
Part 2: Absorption rate constant (Ka) of spironolactone (time^-1) in the multiple-dose period | Pre-dose (Day 1) to 22-26 hours post-dose (Day 11)
  Patients will be assigned to a pharmacokinetic sampling schedule as follows:
  Group 1, Subgroup 1 - Day 1: pre-dose; Day 10; 0.08-0.5 hours, 1-1.5 hours, 2-3 hours, 4-6 hours, 10-13 hours post-dose; Day 11: 22-26 hours post-dose
  Group 1, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.5-1 hour, 1.5-2 hours, 3-4 hours, 6-8 hours post-dose; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 1 - Day 1: pre-dose; Day 10: 0.08-0.75 hours, 1.5-2.5 hours, 3.5-6 hours, 10-13 hours; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.75-1.5 hours, 2.5-3.5 hours, 6-8 hours, 10-13 hours post-dose
  Group 4: the pharmacokinetic sampling schedule during the multiple-dose period for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3.
Part 1: Total clearance from plasma after oral administration (CL/F) of spironolactone in the multiple-dose period | Pre-dose (Day 1) to 22-26 hours post-dose (Day 11)
  Patients will be assigned to a pharmacokinetic sampling schedule as follows:
  Group 1, Subgroup 1 - Day 1: pre-dose; Day 10; 0.08-0.5 hours, 1-1.5 hours, 2-3 hours, 4-6 hours, 10-13 hours post-dose; Day 11: 22-26 hours post-dose
  Group 1, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.5-1 hour, 1.5-2 hours, 3-4 hours, 6-8 hours post-dose; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 1 - Day 1: pre-dose; Day 10: 0.08-0.75 hours, 1.5-2.5 hours, 3.5-6 hours, 10-13 hours; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.75-1.5 hours, 2.5-3.5 hours, 6-8 hours, 10-13 hours post-dose
  Group 4: the pharmacokinetic sampling schedule during the multiple-dose period for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3.
Part 2: Total clearance from plasma after oral administration (CL/F) of spironolactone in the multiple-dose period | Pre-dose (Day 1) to 22-26 hours post-dose (Day 11)
  Patients will be assigned to a pharmacokinetic sampling schedule as follows:
  Group 1, Subgroup 1 - Day 1: pre-dose; Day 10; 0.08-0.5 hours, 1-1.5 hours, 2-3 hours, 4-6 hours, 10-13 hours post-dose; Day 11: 22-26 hours post-dose
  Group 1, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.5-1 hour, 1.5-2 hours, 3-4 hours, 6-8 hours post-dose; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 1 - Day 1: pre-dose; Day 10: 0.08-0.75 hours, 1.5-2.5 hours, 3.5-6 hours, 10-13 hours; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.75-1.5 hours, 2.5-3.5 hours, 6-8 hours, 10-13 hours post-dose
  Group 4: the pharmacokinetic sampling schedule during the multiple-dose period for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3.
Part 1: Volume of distribution after oral administration (V/F) of spironolactone in the multiple-dose period | Pre-dose (Day 1) to 22-26 hours post-dose (Day 11)
  Patients will be assigned to a pharmacokinetic sampling schedule as follows:
  Group 1, Subgroup 1 - Day 1: pre-dose; Day 10; 0.08-0.5 hours, 1-1.5 hours, 2-3 hours, 4-6 hours, 10-13 hours post-dose; Day 11: 22-26 hours post-dose
  Group 1, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.5-1 hour, 1.5-2 hours, 3-4 hours, 6-8 hours post-dose; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 1 - Day 1: pre-dose; Day 10: 0.08-0.75 hours, 1.5-2.5 hours, 3.5-6 hours, 10-13 hours; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.75-1.5 hours, 2.5-3.5 hours, 6-8 hours, 10-13 hours post-dose
  Group 4: the pharmacokinetic sampling schedule during the multiple-dose period for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3.
Part 2: Volume of distribution after oral administration (V/F) of spironolactone in the multiple-dose period | Pre-dose (Day 1) to 22-26 hours post-dose (Day 11)
  Patients will be assigned to a pharmacokinetic sampling schedule as follows:
  Group 1, Subgroup 1 - Day 1: pre-dose; Day 10; 0.08-0.5 hours, 1-1.5 hours, 2-3 hours, 4-6 hours, 10-13 hours post-dose; Day 11: 22-26 hours post-dose
  Group 1, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.5-1 hour, 1.5-2 hours, 3-4 hours, 6-8 hours post-dose; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 1 - Day 1: pre-dose; Day 10: 0.08-0.75 hours, 1.5-2.5 hours, 3.5-6 hours, 10-13 hours; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.75-1.5 hours, 2.5-3.5 hours, 6-8 hours, 10-13 hours post-dose
  Group 4: the pharmacokinetic sampling schedule during the multiple-dose period for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3.
Part 1: Total clearance from plasma after oral administration (CL/F) of canrenone in the multiple-dose period | Pre-dose (Day 1) to 22-26 hours post-dose (Day 11)
  Patients will be assigned to a pharmacokinetic sampling schedule as follows:
  Group 1, Subgroup 1 - Day 1: pre-dose; Day 10; 0.08-0.5 hours, 1-1.5 hours, 2-3 hours, 4-6 hours, 10-13 hours post-dose; Day 11: 22-26 hours post-dose
  Group 1, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.5-1 hour, 1.5-2 hours, 3-4 hours, 6-8 hours post-dose; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 1 - Day 1: pre-dose; Day 10: 0.08-0.75 hours, 1.5-2.5 hours, 3.5-6 hours, 10-13 hours; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.75-1.5 hours, 2.5-3.5 hours, 6-8 hours, 10-13 hours post-dose
  Group 4: the pharmacokinetic sampling schedule during the multiple-dose period for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3.
Part 2: Total clearance from plasma after oral administration (CL/F) of canrenone in the multiple-dose period | Pre-dose (Day 1) to 22-26 hours post-dose (Day 11)
  Patients will be assigned to a pharmacokinetic sampling schedule as follows:
  Group 1, Subgroup 1 - Day 1: pre-dose; Day 10; 0.08-0.5 hours, 1-1.5 hours, 2-3 hours, 4-6 hours, 10-13 hours post-dose; Day 11: 22-26 hours post-dose
  Group 1, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.5-1 hour, 1.5-2 hours, 3-4 hours, 6-8 hours post-dose; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 1 - Day 1: pre-dose; Day 10: 0.08-0.75 hours, 1.5-2.5 hours, 3.5-6 hours, 10-13 hours; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.75-1.5 hours, 2.5-3.5 hours, 6-8 hours, 10-13 hours post-dose
  Group 4: the pharmacokinetic sampling schedule during the multiple-dose period for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3.
Part 1: Volume of distribution after oral administration (V/F) of canrenone in the multiple-dose period | Pre-dose (Day 1) to 22-26 hours post-dose (Day 11)
  Patients will be assigned to a pharmacokinetic sampling schedule as follows:
  Group 1, Subgroup 1 - Day 1: pre-dose; Day 10; 0.08-0.5 hours, 1-1.5 hours, 2-3 hours, 4-6 hours, 10-13 hours post-dose; Day 11: 22-26 hours post-dose
  Group 1, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.5-1 hour, 1.5-2 hours, 3-4 hours, 6-8 hours post-dose; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 1 - Day 1: pre-dose; Day 10: 0.08-0.75 hours, 1.5-2.5 hours, 3.5-6 hours, 10-13 hours; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.75-1.5 hours, 2.5-3.5 hours, 6-8 hours, 10-13 hours post-dose
  Group 4: the pharmacokinetic sampling schedule during the multiple-dose period for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3.
Part 2: Volume of distribution after oral administration (V/F) of canrenone in the multiple-dose period | Pre-dose (Day 1) to 22-26 hours post-dose (Day 11)
  Patients will be assigned to a pharmacokinetic sampling schedule as follows:
  Group 1, Subgroup 1 - Day 1: pre-dose; Day 10; 0.08-0.5 hours, 1-1.5 hours, 2-3 hours, 4-6 hours, 10-13 hours post-dose; Day 11: 22-26 hours post-dose
  Group 1, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.5-1 hour, 1.5-2 hours, 3-4 hours, 6-8 hours post-dose; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 1 - Day 1: pre-dose; Day 10: 0.08-0.75 hours, 1.5-2.5 hours, 3.5-6 hours, 10-13 hours; Day 11: 22-26 hours post-dose
  Groups 2 and 3, Subgroup 2 - Day 1: pre-dose; Day 10: pre-dose, 0.75-1.5 hours, 2.5-3.5 hours, 6-8 hours, 10-13 hours post-dose
  Group 4: the pharmacokinetic sampling schedule during the multiple-dose period for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3.
Part 1: Change from baseline in body weight (kg) (Groups 1 through 3) | Day 1 to Day 18
  Body weight should be measured using the same scale each time and will be reported at: Screening; Day 1: pre-dose (baseline) and anytime between 6 and 8 hours post-dose; Day 5: pre-dose; Day 10: pre-dose and 6 to 8 hours post-dose; Day 11: 22 to 26 hours post-dose; Day 18: during visit.
Part 1: Change from baseline in body weight (kg) (Group 4) | Day 1 to Day 26
  Body weight should be measured using the same scale each time and will be reported at: Screening; Day 1: pre-dose (baseline), and anytime between 6 and 8 hours post-dose; Day 3: anytime between 46 and 50 hours post-dose; Day 8: 166 to 170 hours post-dose; Day 8: 166 to 170 hours post-dose; Day 9: pre-dose and anytime between 6 and 8 hours post-dose; Day 13: pre-dose; Day 18: pre-dose and 6 to 8 hours post-dose; Day 19: 22 to 26 hours post-dose; Day 26: during visit.
Part 2: Change from baseline in body weight (kg) (Groups 1 through 3) | Day 1 to Day 18
  Body weight should be measured using the same scale each time and will be reported at: Screening; Day 1: pre-dose (baseline) and anytime between 6 and 8 hours post-dose; Day 5: pre-dose; Day 10: pre-dose and 6 to 8 hours post-dose; Day 11: 22 to 26 hours post-dose; Day 18: during visit.
Part 2: Change from baseline in body weight (kg) (Group 4) | Day 1 to Day 26
  Body weight should be measured using the same scale each time and will be reported at: Screening; Day 1: pre-dose (baseline), and anytime between 6 and 8 hours post-dose; Day 3: anytime between 46 and 50 hours post-dose; Day 8: 166 to 170 hours post-dose; Day 8: 166 to 170 hours post-dose; Day 9: pre-dose and anytime between 6 and 8 hours post-dose; Day 13: pre-dose; Day 18: pre-dose and 6 to 8 hours post-dose; Day 19: 22 to 26 hours post-dose; Day 26: during visit.
Part 1: Change from baseline in sodium/potassium (Na/K) ratio (Groups 1 through 3) | Day -1 to Day 11
  The Na/K ratio (mmol/mmol) will be calculated using data from spot urine (all groups) and 24-hour urine chemistry (Groups 1 and 2) collection.
  Spot urine will be collected for analysis of electrolytes at the following timepoints in all groups: Day -1: late afternoon/prior to dinner and last void prior to bedtime; Day 1: first morning void; Day 10: late afternoon/prior to dinner and last void prior to bedtime; Day 11: first morning void.
  24-hour urine will be collected for analysis of electrolytes in Groups 1 and 2 only. Urine collection begins on Day -1 AFTER the first morning void and ends AFTER the first morning void on Day 1. Urine collection should start AFTER the first morning void on Day 10 and end AFTER the first morning void on Day 11.
Part 1: Change from baseline in sodium/potassium (Na/K) ratio (Group 4) | Day 8 to Day 19
  The Na/K ratio (mmol/mmol) will be calculated using data from spot urine (all groups) and 24-hour urine chemistry (Groups 1 and 2) collection.
  Spot urine will be collected for analysis of electrolytes at the following timepoints: Day 8: late afternoon/prior to dinner and last void prior to bedtime; Day 9: first morning void; Day 18: late afternoon/prior to dinner and last void prior to bedtime; Day 19: first morning void.
Part 2: Change from baseline in sodium/potassium (Na/K) ratio (Groups 1 through 3) | Day -1 to Day 11
  The Na/K ratio (mmol/mmol) will be calculated using data from spot urine (all groups) and 24-hour urine chemistry (Groups 1 and 2) collection.
  Spot urine will be collected for analysis of electrolytes at the following timepoints in all groups: Day -1: late afternoon/prior to dinner and last void prior to bedtime; Day 1: first morning void; Day 10: late afternoon/prior to dinner and last void prior to bedtime; Day 11: first morning void.
  24-hour urine will be collected for analysis of electrolytes in Groups 1 and 2 only. Urine collection begins on Day -1 AFTER the first morning void and ends AFTER the first morning void on Day 1. Urine collection should start AFTER the first morning void on Day 10 and end AFTER the first morning void on Day 11.
Part 2: Change from baseline in sodium/potassium (Na/K) ratio (Group 4) | Day 8 to Day 19
  The Na/K ratio (mmol/mmol) will be calculated using data from spot urine (all groups) and 24-hour urine chemistry (Groups 1 and 2) collection.
  Spot urine will be collected for analysis of electrolytes at the following timepoints: Day 8: late afternoon/prior to dinner and last void prior to bedtime; Day 9: first morning void; Day 18: late afternoon/prior to dinner and last void prior to bedtime; Day 19: first morning void.
Part 1: Change from baseline in fractional excretion of sodium (FENa; %) (Groups 1 through 3) | Day -1 to Day 11
  FENa will be calculated using data from spot urine (all groups) and 24-hour urine chemistry (Groups 1 and 2) collection.
  Spot urine will be collected for analysis of electrolytes at the following timepoints in all groups: Day -1: late afternoon/prior to dinner and last void prior to bedtime; Day 1: first morning void; Day 10: late afternoon/prior to dinner and last void prior to bedtime; Day 11: first morning void.
  24-hour urine will be collected for analysis of electrolytes in Groups 1 and 2 only. Urine collection begins on Day -1 AFTER the first morning void and ends AFTER the first morning void on Day 1. Urine collection should start AFTER the first morning void on Day 10 and end AFTER the first morning void on Day 11.
  FENa will be calculated as follows:
  [(urine sodium × plasma creatinine)/plasma sodium × urine creatinine) × 100]
Part 1: Change from baseline in fractional excretion of sodium (FENa; %) (Group 4) | Day 8 to Day 19
  FENa will be calculated using data from spot urine (all groups) and 24-hour urine chemistry (Groups 1 and 2) collection.
  Spot urine will be collected for analysis of electrolytes at the following timepoints: Day 8: late afternoon/prior to dinner and last void prior to bedtime; Day 9: first morning void; Day 18: late afternoon/prior to dinner and last void prior to bedtime; Day 19: first morning void.
  FENa will be calculated as follows:
  [(urine sodium × plasma creatinine)/plasma sodium × urine creatinine) × 100]
Part 2: Change from baseline in fractional excretion of sodium (FENa; %) (Groups 1 through 3) | Day -1 to Day 11
  FENa will be calculated using data from spot urine (all groups) and 24-hour urine chemistry (Groups 1 and 2) collection.
  Spot urine will be collected for analysis of electrolytes at the following timepoints in all groups: Day -1: late afternoon/prior to dinner and last void prior to bedtime; Day 1: first morning void; Day 10: late afternoon/prior to dinner and last void prior to bedtime; Day 11: first morning void.
  24-hour urine will be collected for analysis of electrolytes in Groups 1 and 2 only. Urine collection begins on Day -1 AFTER the first morning void and ends AFTER the first morning void on Day 1. Urine collection should start AFTER the first morning void on Day 10 and end AFTER the first morning void on Day 11.
  FENa will be calculated as follows:
  [(urine sodium × plasma creatinine)/plasma sodium × urine creatinine) × 100]
Part 2: Change from baseline in fractional excretion of sodium (FENa; %) (Group 4) | Day 8 to Day 19
  FENa will be calculated using data from spot urine (all groups) and 24-hour urine chemistry (Groups 1 and 2) collection.
  Spot urine will be collected for analysis of electrolytes at the following timepoints: Day 8: late afternoon/prior to dinner and last void prior to bedtime; Day 9: first morning void; Day 18: late afternoon/prior to dinner and last void prior to bedtime; Day 19: first morning void.
  FENa will be calculated as follows:
  [(urine sodium × plasma creatinine)/plasma sodium × urine creatinine) × 100]

SECONDARY OUTCOMES:
Parts 1 and 2: Incidence of adverse events, serious adverse events, and adverse events leading to discontinuation during the single-dose periods (Group 4 only) | Day 1 to Day 8
Parts 1 and 2: Number of patients with clinically significant findings from clinical laboratory tests, vital signs, and physical examinations during the single-dose periods (Group 4 only) | Day 1 to Day 8
Parts 1 and 2: Absorption rate constant (Ka) of spironolactone (time^-1) in the single-dose period (Group 4 only) | Day 1 to Day 8
  The pharmacokinetic sampling schedule for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3, but samples will likely be collected on Days 1, 3, and 8. The number of PK samples collected may be reduced from this preliminary schedule based on review of PK concentration-time data from Groups 1 to 3 and will not exceed allowable limits for blood volume collection in neonates and infants in 1 day and within 30 days.
Parts 1 and 2: Total clearance from plasma after oral administration (CL/F) of spironolactone in the single-dose period (Group 4 only) | Day 1 to Day 8
  The pharmacokinetic sampling schedule for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3, but samples will likely be collected on Days 1, 3, and 8. The number of PK samples collected may be reduced from this preliminary schedule based on review of PK concentration-time data from Groups 1 to 3 and will not exceed allowable limits for blood volume collection in neonates and infants in 1 day and within 30 days.
Parts 1 and 2: Volume of distribution after oral administration (V/F) of spironolactone in the single-dose period (Group 4 only) | Day 1 to Day 8
  The pharmacokinetic sampling schedule for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3, but samples will likely be collected on Days 1, 3, and 8. The number of PK samples collected may be reduced from this preliminary schedule based on review of PK concentration-time data from Groups 1 to 3 and will not exceed allowable limits for blood volume collection in neonates and infants in 1 day and within 30 days.
Parts 1 and 2: Total clearance from plasma after oral administration (CL/F) of canrenone in the single-dose period (Group 4 only) | Day 1 to Day 8
  The pharmacokinetic sampling schedule for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3, but samples will likely be collected on Days 1, 3, and 8. The number of PK samples collected may be reduced from this preliminary schedule based on review of PK concentration-time data from Groups 1 to 3 and will not exceed allowable limits for blood volume collection in neonates and infants in 1 day and within 30 days.
Parts 1 and 2: Volume of distribution after oral administration (V/F) of canrenone in the single-dose period (Group 4 only) | Day 1 to Day 8
  The pharmacokinetic sampling schedule for Group 4 will be determined following Safety Review Committee of data from Groups 1 through 3, but samples will likely be collected on Days 1, 3, and 8. The number of PK samples collected may be reduced from this preliminary schedule based on review of PK concentration-time data from Groups 1 to 3 and will not exceed allowable limits for blood volume collection in neonates and infants in 1 day and within 30 days.
Part 1: Incidence of adverse events, serious adverse events, and adverse events leading to discontinuation during the multiple-dose period (Groups 1 through 3) | Day 1 to Day 41
Part 1: Incidence of adverse events, serious adverse events, and adverse events leading to discontinuation during the multiple-dose period (Group 4 only) | Day 9 to Day 49
Part 2: Incidence of adverse events, serious adverse events, and adverse events leading to discontinuation during the multiple-dose period (Groups 1 through 3) | Day 1 to Day 41
Part 2: Incidence of adverse events, serious adverse events, and adverse events leading to discontinuation during the multiple-dose period (Group 4 only) | Day 9 to Day 49
Part 1: Number of patients with clinically significant findings from clinical laboratory tests, vital signs, and physical examinations during the multiple-dose period (Groups 1 through 3) | Day 1 to Day 41
Part 1: Number of patients with clinically significant findings from clinical laboratory tests, vital signs, and physical examinations during the multiple-dose period (Group 4 only) | Day 9 to Day 49
Part 2: Number of patients with clinically significant findings from clinical laboratory tests, vital signs, and physical examinations during the multiple-dose period (Groups 1 through 3) | Day 1 to Day 41
Part 2: Number of patients with clinically significant findings from clinical laboratory tests, vital signs, and physical examinations during the multiple-dose period (Group 4 only) | Day 9 to Day 49
Part 1: Change from baseline in abdominal girth (cm) (Groups 1 through 3) | Day 1 to Day 10
  Abdominal girth is the measurement of the distance around the abdomen at a specific point, usually the level of the navel, and will be measured on Day 1: pre-dose; Day 5: pre-dose; and Day 10: pre-dose.
Part 1: Change from baseline in abdominal girth (cm) (Group 4) | Day 8 to Day 18
  Abdominal girth is the measurement of the distance around the abdomen at a specific point, usually the level of the navel, and will be measured on Day 8: 166 to 170 h post-dose; Day 9: pre-dose; Day 13: pre-dose; Day 18: pre-dose.
Part 2: Change from baseline in abdominal girth (cm) (Groups 1 through 3) | Day 1 to Day 10
  Abdominal girth is the measurement of the distance around the abdomen at a specific point, usually the level of the navel, and will be measured on Day 1: pre-dose; Day 5: pre-dose; and Day 10: pre-dose.
Part 2: Change from baseline in abdominal girth (cm) (Group 4) | Day 8 to Day 18
  Abdominal girth is the measurement of the distance around the abdomen at a specific point, usually the level of the navel, and will be measured on Day 8: 166 to 170 h post-dose; Day 9: pre-dose; Day 13: pre-dose; Day 18: pre-dose.
Part 1: Number of patients with clinically significant findings from electrolytes and other laboratory results (Groups 1 through 3) | Day 1 to Day 18
  Laboratory test results will include serum sodium, potassium, magnesium, blood urea nitrogen, serum creatinine, glycemia, albumin, total proteins, estimated glomerular filtration rate, urinary sodium and potassium, creatinine, and osmolality.
Part 1: Number of patients with clinically significant findings from electrolytes and other laboratory results (Group 4) | Day 9 to Day 26
  Laboratory test results will include serum sodium, potassium, magnesium, blood urea nitrogen, serum creatinine, glycemia, albumin, total proteins, estimated glomerular filtration rate, urinary sodium and potassium, creatinine, and osmolality.
Part 2: Number of patients with clinically significant findings from electrolytes and other laboratory results (Groups 1 through 3) | Day 1 to Day 18
  Laboratory test results will include serum sodium, potassium, magnesium, blood urea nitrogen, serum creatinine, glycemia, albumin, total proteins, estimated glomerular filtration rate, urinary sodium and potassium, creatinine, and osmolality.
Part 2: Number of patients with clinically significant findings from electrolytes and other laboratory results (Group 4) | Day 9 to Day 26
  Laboratory test results will include serum sodium, potassium, magnesium, blood urea nitrogen, serum creatinine, glycemia, albumin, total proteins, estimated glomerular filtration rate, urinary sodium and potassium, creatinine, and osmolality.
Part 1: Levels of N-terminal pro B-type natriuretic peptide (pg/mL) in Groups 1 to 3 | Day 11
Part 1: Levels of N-terminal pro B-type natriuretic peptide (pg/mL) in Group 4 | Day 19
Part 2: Levels of N-terminal pro B-type natriuretic peptide (pg/mL) in Groups 1 to 3 | Day 11
Part 2: Levels of N-terminal pro B-type natriuretic peptide (pg/mL) in Group 4 | Day 19
Part 1: Levels of cystatin C (mg/L) in Groups 1 to 3 | Day 11
Part 1: Levels of cystatin C (mg/L) in Group 4 | Day 19
Part 2: Levels of cystatin C (mg/L) in Groups 1 to 3 | Day 11
Part 2: Levels of cystatin C (mg/L) in Group 4 | Day 19

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Sakowski, Study Director — CMP Pharma